CLINICAL TRIAL: NCT01181284
Title: Modulating Effects of Lisinopril on Sildenafil Activity in PAH (MELISSA)
Brief Title: Modulating Effects of Lisinopril on Sildenafil Activity in Pulmonary Arterial Hypertension(PAH)( MELISSA)
Acronym: MELISSA
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert P. Frantz, MD, Mayo Clinic
Other Study IDs: 08-001716; MELISSA
Record Dates: First submitted 2010-01-07; First posted 2010-08-13 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension (PAH)
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lisinopril: Participants will be randomized 2 to 1 to receive drug versus placebo.

SUMMARY:
Patients with pulmonary arterial hypertension(PAH) suffer from chronic shortness of breath, and have impaired survival related to progressive right ventricular failure. Abnormal vasoreactivity to nitric oxide(NO) plays a role in the pathophysiology of PAH. Phosphodiesterase Type 5 Inhibitor (PDE5 inhibitors) sildenafil have been shown to be beneficial in PAH, but extent of benefit is variable.

DETAILED DESCRIPTION:
The broad aim of this investigation is to determine whether the modulating effect of angiotensin converting enzyme inhibition on vascular smooth muscle responsiveness to the nitric oxide pathway that we have observed in an animal model of Congestive Heart Failure(CHF) can be exploited in humans with PAH. Furthermore, we have identified a group of genes TAO kinase I, IL-10, Rho kinase, Raf1, bile acid coenzyme A and Fmr1 that are modulated by long-acting angiotensin-converting enzyme inhibitor (ACEI) in our animal model, and therefore may also be modulated by ACEI in patients with PAH

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* World Health Organization (WHO) Group I PAH with prior documentation of peripheral vascular resistance (PVR) > 3 WU and wedge(PCW) 16 or less.
* WHO Functional Class I-III
* 6 minute walk distance 150-575 meters
* Women of child bearing potential must have a negative pregnancy test and be using effective contraception
* Receiving therapy with phosphodiesterase-5 inhibitor for PAH (sildenafil or tadalafil) for at least 3 months and with stable dose for at least 30 days
* If already receiving therapy with endothelin receptor antagonists must have been on therapy for at least 3 months and on stable dose for at least 30 days

Exclusion Criteria:

* Allergy or intolerance to captopril or other angiotensin converting enzyme inhibitors
* Systemic systolic blood pressure less than 100 mm Hg
* Therapy with prostanoids (iloprost, treprostinil, epoprostenol) within preceding 3 months
* Pregnant or breast feeding
* Creatinine > 2.0 mg/dl
* Potassium > 5.0 meq/dl
* Unable to provide informed consent
* TLC or VC <60% predicted
* Untreated obstructive sleep apnea
* LVEF < 40%
* Hb < 10 mg/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be currently diagnosed with Pulmonary Arterial Hypertension (PAH). Lisinopril versus placebo will be added to participants already recieving a stable dose of Sildenafil.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The primary aim of the pilot study is to assess feasibility and tolerability. | 32 weeks

SECONDARY OUTCOMES:
Demonstrate tolerability of long-acting angiotensin-converting enzyme inhibitor (ACEI) therapy in this patient cohort | 32 weeks
Demonstrate whether long-acting angiotensin-converting enzyme inhibitor (ACEI) in Pulmonary Arterial Hypertension (PAH) pts on sildenafil modifies regulation of the genes. | 32 weeks
Demonstrate whether ACEI in PAH pts on sildenafil reduces N-BNP levels, a marker of disease severity | 32 weeks
Demonstrate whether ACEI in PAH pts on sildenafil has an effect on pulmonary gas exchange parameters (exhaled NO, Dm, Vc, DLCO). | 32 weeks
Obtain exploratory data regarding whether ACEI in PAH pts on sildenafil improves functional class and 6 minute walk distance. | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Frantz, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States